CLINICAL TRIAL: NCT06261008
Title: Utilization of a Theory-driven, Culturally Tailored, Social Media-based, Interactive Telehealth Intervention to Increase Longitudinal Adherence to Repeat Faecal Immunochemical Test Screening: A Randomized Controlled Trial
Brief Title: Interactive Telehealth Intervention to Increase Longitudinal Adherence to Repeat Faecal Immunochemical Test Screening
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Thomas Yuen Tung Lam, Assistant professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023.553
Record Dates: First submitted 2023-12-04; First posted 2024-02-15 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: CRC, Colorectal Cancer
Keywords: colorectal cancer, screening, fecal immunochemical test
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Patient will be randomized into either standard care or telehealth intervention group
Masking Description: There will no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): An automated noninteractive short message service (SMS) text reminder, used by the Program as standard care (SC), is delivered to participants who are due for repeat FIT.
- Telehealth Intervention group (Experimental): Subjects randomized to the Telehealth Intervention (TI) group will receive the SC as well as an interactive TI with interactive health education messages via a WhatsApp-based chatbot on the repeat FIT due date. All subjects will be followed up on WhatsApp at 3 months after their repeat FIT due date and asked about their repeat FIT status.
  Interventions: Behavioral: TI group

INTERVENTIONS:
Behavioral: TI group — CRC screening is arranged by referring the participants to the government-subsidized population-based CRC screening program. Our center is a PCP clinic offering FIT screenings under the Program. Colonoscopy is arranged if the FIT result is positive. Participants are instructed to repeat FIT at any PCP clinic 2 years after receiving a negative result. Based on the 34% local FIT screening adherence rate under SC and the assumption of improved FIT adherence to 49% after interactive TI, a minimum sample size of 332 subjects (166 per group) is required to achieve a statistical significance of p<0.05 and power of 80%. Assuming that 10% of the subjects will drop out, be lost to follow-up, or have incomplete chatbot conversations, the required sample size is rounded up to 370 (185 per group)
  Arms: Telehealth Intervention group

SUMMARY:
In Hong Kong, Colorectal cancer ranks second in both cancer incidence and mortality. The government-subsidized population-based CRC screening program (the Program) was launched for asymptomatic individuals aged 50-75 years to undergo biennial FIT screenings. A subsidized follow-up colonoscopy is offered to participants with positive FIT results. Participants are advised to repeat the FIT screening 2 years after receiving a negative result. An automated noninteractive short message service (SMS) text reminder, used by the Program as standard care (SC), is delivered to participants who are due for repeat FIT. According to unpublished data, despite SC, only 34% of participants adhere to biennial repeat FIT in the CRC screening program. Nonadherence to repeat FIT screening is caused by forgetfulness and is associated with an individual's psychological health behaviour.

DETAILED DESCRIPTION:
Eligible subject will be randomised to either the TI group or SC group. All subjects will receive an automated SMS text reminder delivered by the Program as the standard care.

Subjects randomized to the TI group will receive the SC as well as an interactive TI with interactive health education messages via a WhatsApp-based chatbot on the repeat FIT due date. All subjects will be followed up on WhatsApp at 3 months after their repeat FIT due date and asked about their repeat FIT status.

Subjects will be invited to participate in four focus group discussions to elucidate how the study intervention influences repeat FIT adherence behaviours, explore the complexity of regular FIT screening, and reveal, based on the participants' accounts, the barriers to and facilitators of their adherence to the repeat FIT screening. The discussion will be audiotaped.

ELIGIBILITY:
Inclusion Criteria:

* 50-75 years old
* already enrolled in the Program with negative FIT results in 2022
* eligible for the Program inclusion and due for repeat FIT screening in 2024
* either the participants themselves or their family members / caregivers have access to and agree to be contacted via WhatsApp
* ability to understand Chinese

Exclusion Criteria:

* who have incomplete conversations with the chatbot, lack of access to WhatsApp, or are unable to provide informed consent will be excluded

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-03-26 (Estimated); Study Completion 2026-06-26 (Estimated)

PRIMARY OUTCOMES:
adherence rate | 3 months
  The primary outcome will be the repeat FIT screening adherence rate defined as returning completed FIT kits within 3 months after the repeat FIT due date in 2024.

SECONDARY OUTCOMES:
the number of days to repeat FIT | 6 months
  the number of days to participate in (FIT kits collection date to intervention date) and complete the repeat FIT screening after the intervention (completed FIT kits return date to intervention date)
costs incurred in each study arm | 6 months
  including the cost of chatbot development, video production and the standard care of SMS reminder
uptake rate in positive FIT | 12 months
  For those who have positive FIT, we will also assess their uptake rate of colonoscopy following positive FIT
detection rate in positive FIT | 12 months
  For those who have positive FIT, we will also assess the detection rate of advanced neoplasm as defined as at least one colorectal cancer or advanced adenoma (size ≥10 mm, tubulovillous or villous component, or high-grade dysplasia).
qualitative factors associated with repeat FIT adherence | 12 months
  Subjects will be invited to join the focus group for assessing qualitative factors associated with repeat FIT adherence in the biennial population-based CRC screening program

CONTACTS AND LOCATIONS:
Locations (1):
- Centre of Digestive Health, Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
There will be no plan to share IPD